CLINICAL TRIAL: NCT01081002
Title: Study of Propofol Sedation During Upper Endoscopy With and Without Topical Pharyngeal Anesthesia
Brief Title: Propofol Sedation During Upper Endoscopy With and Without Topical Pharyngeal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Lukas Degen, Prof., University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EKBB 101/09
Record Dates: First submitted 2010-03-02; First posted 2010-03-05 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2010-03

CONDITIONS: Conscious Sedation
Keywords: Propofol; Conscious sedation; Topical pharyngeal anesthesia; Anesthetics, Local; Gastrointestinal Endoscopy
MeSH Terms: interventions — Lidocaine; gentian root extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anesthesia (=A) with lidocaine 10% (Active Comparator): 3 min before sedation 4 puffs of terbutaline diluted lidocaine solution (Xylocaine ® 10% spray, Astra Zeneca, London, UK) will be sprayed on the pharynx
  Interventions: Drug: Lidocaine 10%
- A with diluted gentian root solution (Placebo Comparator): 3 min before sedation 4 puffs of highly diluted gentian solution will be sprayed on the pharynx
  Interventions: Drug: Diluted gentian root solution

INTERVENTIONS:
Drug: Lidocaine 10% — 3 min before the endoscopy under propofol sedation 4 puffs of lidocaine 10% will be sprayed on the pharynx as a pharyngeal anesthesia
  Other Names: Xylocaine 10% spray
  Arms: Anesthesia (=A) with lidocaine 10%
Drug: Diluted gentian root solution — As a basis, an infusion of water (45%), ethanol (35%) and gentian root cut will be used. The gentian root infusion is approved as a natural flavor in the food industry.3 min before the endoscopy under propofol sedation 4 puffs of this gentian root infusion will be sprayed on the pharynx as a pharyngeal anesthesia
  Other Names: Gentian root extract, CAS no. 72968-42-4
  Arms: A with diluted gentian root solution

SUMMARY:
It is unclear whether a topical pharyngeal anesthesia adds any benefit to the upper gastrointestinal endoscopy under a propofol sedation. We hypothesize that a topical pharyngeal anesthesia does not ease the upper gastrointestinal endoscopy under propofol sedation. The aim of this study is therefore to quantify the impact of a topical pharyngeal anesthesia to the upper gastrointestinal endoscopy in patients sedated with propofol.

Patients will be randomized to receive a topical pharyngeal spray containing either an anesthetic drug (lidocaine 10%) or a placebo. Thereafter the upper endoscopy will be conducted in its standard manner.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled diagnostic upper endoscopy
* Wish to be sedated
* ASA class I - III
* Signed informed consent

Exclusion Criteria:

* Emergency medical examinations
* Therapeutic Endoscopy
* ASA class IV
* Pregnancy
* Known allergy to propofol or lidocaine

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Number triggered gag reflex during the intubation of the endoscope | Start of the exam until the successful intubation of the esophagus with the endoscope
Number of attempts of intubation with the endoscope through the upper esophageal sphincter | Start of the exam until the successful intubation of the esophagus with the endoscope
Extent of salivation during intubation | Start of the exam until the successful intubation of the esophagus with the endoscope

SECONDARY OUTCOMES:
Amount of propofol used to successfully intubate the esophagus | Start of the exam until the successful intubation of the esophagus with the endoscope
Total amount of propofol used during the investigation | From the start until the end of the exam
Overall assessment of the procedure by the endoscopist | Immediately after finishing the endoscopy
Assumption of the endoscopist if lidocaine or placebo has been used | Immediately after finishing the endoscopy
Overall assessment of the investigation by the patient | Immediately after recovery of consciousness of the patient
Extent of amnesia in the patient | Immediately after recovery of consciousness of the patient
Experienced problems (aspiration, bronchospasm, desaturation) | From the start until the end of the exam
The impact of the individual endoscopists or registered nurses involved in the endoscopy | After finishing the entire study

CONTACTS AND LOCATIONS:
Overall Officials: Ludwig T Heuss, MD, Principal Investigator — Spital Zollikerberg; Lukas Degen, Prof, Principal Investigator — University Hospital, Basel, Switzerland
Locations (2):
- Switzerland (2):
  - University Hospital; Division of Gastroenterology and Hepatology, Basel, Canton of Basel-City
  - Hospital of Zollikerberg, Internal Medicine, Zollikerberg, Canton of Zurich

REFERENCES:
- [Derived] Heuss LT, Hanhart A, Dell-Kuster S, Zdrnja K, Ortmann M, Beglinger C, Bucher HC, Degen L. Propofol sedation alone or in combination with pharyngeal lidocaine anesthesia for routine upper GI endoscopy: a randomized, double-blind, placebo-controlled, non-inferiority trial. Gastrointest Endosc. 2011 Dec;74(6):1207-14. doi: 10.1016/j.gie.2011.07.072. Epub 2011 Oct 13. PMID 22000794